CLINICAL TRIAL: NCT07386873
Title: Randomized Controlled Trial on the Efficacy of Olfactory Cleft Steroid Drops in Patients With Chronic Rhinosinusitis With Olfactory Cleft Obstruction
Brief Title: The Efficacy of Olfactory Cleft Steroid Drops in Patients With CRS With Olfactory Cleft Obstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9059107
Record Dates: First submitted 2026-01-24; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis (CRS); Smell Dysfunction
Keywords: Olfactory dysfunction; Chronic rhinosinusitis; Steroid nasal drops; Olfactory cleft obstruction
MeSH Terms: conditions — Olfaction Disorders | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Drops Group (Experimental)
  Interventions: Device: Nasal Drops
- Standard Nasal Spray Group (Active Comparator)
  Interventions: Device: Nasal Spray

INTERVENTIONS:
Device: Nasal Drops — Patients will assume the Mygind position (supine with head extended over the edge of the bed, nostrils facing upward). Five drops of budesonide suspension (2ml:1mg) will be administered into each nostril to ensure delivery to the olfactory cleft at the nasal apex. The position will be maintained for approximately 5 minutes, after which any residual medication in the oral or nasal cavity may be expelled. This procedure will be performed twice daily (morning and evening) for 3 months. During the first month, olfactory function will be assessed weekly, with a nasal sinus CT scan at the end of the month. In the second month, olfactory evaluations will be conducted biweekly, followed by a final assessment at the end of the third month.
  Arms: Nasal Drops Group
Device: Nasal Spray — Patients will use budesonide nasal spray administered in the same Mygind position, with 2 sprays per nostril (total daily dose: 200μg). After administration, patients will gently sniff to facilitate drug dispersion. The treatment duration and follow-up schedule will be identical to the experimental group.
  Arms: Standard Nasal Spray Group

SUMMARY:
This study aims to compare the efficacy of steroid nasal drops targeting the olfactory cleft versus traditional intranasal steroid sprays in improving olfactory function in patients with chronic rhinosinusitis (CRS) with olfactory cleft obstruction. The main questions this clinical trial aims to answer are:

1. Efficacy Comparison: Is olfactory improvement greater with olfactory cleft-targeted steroid nasal drops compared to standard nasal steroid sprays in CRS patients?
2. Mechanism Exploration: How do changes in inflammatory markers, obstruction severity, and olfactory test results explain the potential benefits of this treatment approach?

DETAILED DESCRIPTION:
Olfactory dysfunction is one of the most common clinical symptoms in patients with chronic rhinosinusitis (CRS), affecting approximately 60%-80% of individuals with CRS. This condition significantly impairs quality of life and is associated with systemic health issues such as depression and nutritional imbalances. The olfactory cleft, a critical anatomical region housing the olfactory neuroepithelium, is often obstructed in CRS patients due to nasal polyps or mucosal hypertrophy, leading to conductive olfactory dysfunction.

Current first-line treatments for CRS, including oral or intranasal corticosteroids, have limitations. Oral steroids pose systemic side effects, while standard nasal sprays often fail to deliver adequate drug concentrations to the olfactory cleft. In contrast, targeted hormone nasal drops may achieve higher efficacy by directly addressing localized inflammation and edema in the olfactory cleft. Preliminary studies suggest that fluticasone nasal drops can reduce the need for sinus surgery in patients with CRS unresponsive to conventional sprays. However, no randomized controlled trials have systematically evaluated the efficacy of olfactory cleft-targeted hormone drops in improving olfactory function in CRS patients with confirmed olfactory cleft obstruction.

In this study, investigators planned to enroll 54 patients with olfactory cleft obstruction and assign them to one of two treatments: olfactory cleft-targeted steroid nasal drops or conventional nasal sprays. This study aims to investigate the efficacy and underlying mechanisms of olfactory cleft-targeted steroid nasal drops in improving olfactory function.

ELIGIBILITY:
Inclusion Criteria:

1. Prospective enrollment of otolaryngology clinic patients aged 18-65 years with olfactory dysfunction. Diagnosis of chronic rhinosinusitis-related olfactory dysfunction is based on the EPOS 2020 guidelines. Participants must demonstrate olfactory impairment via Sniffin' Sticks testing, with TDI scores (sum of Threshold, Discrimination, and Identification) meeting:(1) Hyposmia: 16 < TDI < 30.75; (2) 3.Anosmia: TDI < 15.
2. Sinus CT scans confirming obstruction in the olfactory cleft region.
3. Willingness to participate and signed informed consent.

Exclusion Criteria:

1. Use of systemic corticosteroids within 4 weeks or intranasal steroids within 2 weeks prior to enrollment.
2. Severe nasal septum deviation, nasal tumors, acute upper respiratory infections, or uncontrolled allergic rhinitis.
3. Severe cardiovascular disease, hepatic/renal insufficiency, uncontrolled diabetes, or immune system disorders.
4. Current or planned pregnancy.
5. Investigator-determined inability to comply with study requirements (e.g., memory/behavioral disorders, depression, heavy alcohol use, prior non-compliance).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Sniffin' Sticks test | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  A clinically significant olfactory improvement as measured by Sniffin' Sticks threshold, discrimination, and identification(TDI)

SECONDARY OUTCOMES:
Subjective Olfactory Improvement and Nasal Symptoms | 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  Patient-reported olfactory improvement measured using the Olfactory-Visual Analogue Scale (VAS) and nasal symptoms assessed via the the Sino-Nasal Outcome Test 22 (SNOT-22) questionnaire. These measures evaluate treatment effects on self-perceived smell recovery and associated nasal complaints.
CT Evaluation of Olfactory Cleft Blockage | Baseline and 4 weeks after the initiation of treatment.
Inflammatory Marker Levels in Olfactory Mucosa | Baseline and 4 weeks after the initiation of treatment.
  Analysis of inflammatory cytokines via ELISA and single-cell sequencing from olfactory mucosal brush samples, with concurrent serum inflammatory marker testing.
Adverse Event | 1 week, and 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks after the initiation of treatment.
  Documentation of local (nasal irritation, epistaxis) and systemic steroid-related adverse events using standardized case report forms during all follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Dawei Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.